CLINICAL TRIAL: NCT06698211
Title: Evaluation of Posaconazole Tablet As Primary Prophylaxis of Hematopoietic Stem Cell Transplant Patients with Gastrointestinal GVHD
Brief Title: Posaconazole Tablet As Primary Prophylaxis of HSCT Patients with Gastrointestinal GVHD
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2024039
Record Dates: First submitted 2024-10-23; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Invasive Fungal Disease; Graft Versus Host Disease; Hematopoietic Stem Cell Transplantation
Keywords: hematopoietic stem cell transplantation; graft versus host disease; invasive fungal disease; primary prophylaxis
MeSH Terms: conditions — Invasive Fungal Infections; Graft vs Host Disease | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Posaconazole tablet: Posaconazole tablet will be given at a dose of 300mg q12h on day 1 and 300mg qd from day 2 for patients who receive HSCT as the primary prophylaxis of IFD, after which the Posaconazole plasma concentration on day 5 will be examined.
  Interventions: Drug: Posaconazole tablet

INTERVENTIONS:
Drug: Posaconazole tablet — Posaconazole tablet will be given at a dose of 300mg q12h on day 1 and 300mg qd from day 2 for patients who receive HSCT as the primary prophylaxis of IFD, after which the Posaconazole plasma concentration on day 5 will be examined. Once patients developed GI GVHD, first line therapy and second line treatment will be reviewed according to the condition, besides which the Posaconazole plasma concentration would be detected again on the first, third and fifth day after onset of GI GVHD symptoms to monitor the impact of GI GVHD on the Posaconazole plasma concentration.

SUMMARY:
This is a prospective investigation using a nonrandomized, single-arm design. Posaconazole tablet will be given at a dose of 300mg q12h on day 1 and 300mg qd from day 2 for patients who receive HSCT as the primary prophylaxis of IFD, after which the Posaconazole plasma concentration on day 5 will be examined.

DETAILED DESCRIPTION:
This is a prospective investigation using a nonrandomized, single-arm design. Posaconazole tablet will be given at a dose of 300mg q12h on day 1 and 300mg qd from day 2 for patients who receive HSCT as the primary prophylaxis of IFD, after which the Posaconazole plasma concentration on day 5 will be examined. Once patients developed GI GVHD, first line therapy and second line treatment will be reviewed according to the condition, besides which the Posaconazole plasma concentration would be detected again on the first, third and fifth day after onset of GI GVHD symptoms to monitor the impact of GI GVHD on the Posaconazole plasma concentration. The primary endpoint was the incidence of breakthrough fungal infection (BFI) including proven, probable and possible fungal infection

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic diseases who undergoes hematopoietic stem cell transplantation.
2. Patients who receive Posaconazole tablet as primary prophylaxis of invasive fungal disease.
3. Patients developing or developed acute gastrointestinal GVHD which require systemic immunosuppressive therapy of corticosteroids with- or-without other immunosuppressive agents including calcineurin inhibitors.

   Gastrointestinal GVHD grades (I-IV) were recorded according to the Glucksberg criteria.
4. Patients themselves or their authorized clients agree to participate in the clinical study and sign the informed consent

Exclusion Criteria:

1. refuse to enroll
2. patients have known hypersensitivity or other serious adverse reaction to any azole antifungal therapy, or to any other ingredient of the study medication used.
3. pregnant or lactating females
4. take drugs known to interfere with azole antifungal agents, including terfenadine, cisapride and ebastine, within 24h before Posaconazole application; astemizole at enrollment or within 10 days before Posaconazole application; or cimetidine, rifampin, carbamazepine, phenytoin, rifamycin, barbiturates, isoniazid, catharanthine and anthracyclines within 24 h before Posaconazole application
5. have an ECG with a prolonged QTc interval (QTc greater than 500 ms);
6. have severe renal insufficiency, alanine transaminase, aspartate transaminase, alkaline phosphatase or total bilirubin levels more than two-times the upper limit of normal;
7. patients are expected to survive no more than 72 h;
8. Those with evidence of active fungal infection within 3 weeks prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patient undergoing Hematopoietic stem cell transplantation who meet the inclusion criteria and do not meet the exclusion criteria can enroll in this study.
  2. Ages eligible for study: 18-75
  3. Sexes eligible for study: All
  4. Race: Chinese
  5. Ethnicity: All
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
primary endpoint | From 7 days after starting posaconazole prophylaxis post-transplant to 7 days after the end of prophylaxis
  1. The incidence of breakthrough fungal infection (BFI) including proven, probable and possible fungal infection

SECONDARY OUTCOMES:
2 | Day 5 after posaconazole administration, and Days 1, 3, and 7 after the onset of gastrointestinal GVHD
  Posaconazole plasma concentration
3 | From the first day of posaconazole prophylaxis for IFD post-transplant to the end of prophylaxis.
  Gastrointestinal GVHD grade, diarrhea status (frequency, volume), use and adjustment of immunosuppressants, neutrophil count
4 | From the first day of posaconazole prophylaxis for IFD post-transplant to the end of prophylaxis.
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Pang, doctor, Principal Investigator — Hematopoietic stem cell transplantation Center
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
Data sharing is not considered for the time being due to patient privacy concerns.